CLINICAL TRIAL: NCT06014632
Title: The Effect of Supervised Motor Control Exercise Program on Pain, Disability, Kinesiophobia, Proprioception and Function After Lumbar Spinal Decompression Surgery
Brief Title: Efficacy of Motor Control Exercise Program After Lumbar Spinal Decompression Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Muğla Sıtkı Koçman University (Other)
Responsible Party: Principal Investigator, Fatih Ozden, Assistant Professor, Muğla Sıtkı Koçman University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NRŞ RKÇ
Record Dates: First submitted 2023-08-17; First posted 2023-08-28 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Lumbar Spine Disease
MeSH Terms: conditions — Spinal Diseases | interventions — Rehabilitation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): The study group will be given motor control exercises in addition to the program given to the control group. It will include exercise therapy aimed at improving the motor control of the lumbar spine. These applications will be applied to the patients face-to-face in a clinical setting 2 days a week for 12 weeks. In addition, both groups will be told that they can contact the researcher upon request.
  Interventions: Other: Rehabilitation
- Control Group (Active Comparator): The control group will receive stretching, strengthening, core stabilization and educational content as usual care.
  Interventions: Other: Control

INTERVENTIONS:
Other: Rehabilitation — The study group will be given motor control exercises in addition to the program given to the control group.
  Arms: Intervention Group
Other: Control — The control group will receive stretching, strengthening, core stabilization and educational content as usual care.
  Arms: Control Group

SUMMARY:
The study will be conducted with volunteer patients who have undergone lumbar decompression surgery and who are followed up by the Neurosurgery outpatient clinic of Fethiye State Hospital. The cases will be divided into 2 groups by randomization software. The control group will receive stretching, strengthening, core stabilization and educational content as usual care 3 months post-operatively. The study group will be given motion control exercises in addition to the program given to the control group 3 months post-operatively. These applications will be applied to the patients face-to-face in the clinical environment 2 days a week for 12 weeks. The first evaluation will be performed 3 months post-operatively before the treatment and the second evaluation will be performed 3 months after the treatment.

ELIGIBILITY:
Inclusion Criteria:

* To have undergone lumbar decompression surgery without fusion and 3 months have passed, to participate in all necessary follow-up evaluations and treatment sessions
* To be between the ages of 18-65, to be able to understand simple commands and to have signed the consent form

Exclusion Criteria:

* Presence of a previous spinal fusion surgery, presence of malignancy
* Having undergone spine surgery before
* Have any other orthopedic or neurological problem that may affect treatment and assessments
* Situations that may interfere with communication
* Lack of cooperation during the study and refusal to participate in the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2023-06-12 (Actual); Primary Completion 2025-09-01 (Actual); Study Completion 2025-12-01 (Actual)

PRIMARY OUTCOMES:
12-item Örebro Musculoskeletal Screening Questionnaire (ÖMSQ-12) | Change from Baseline ÖMSQ-12 at 12 weeks
  ÖMSQ-12 is a 12-item self-report questionnaire. Each item is scored on an 11-point Likert scale (0-10) based on the response to the question asked. Items 8, 11 and 12 are reverse scored items. The maximum score that can be obtained from the questionnaire is 120. A high score means a high risk of absenteeism, high cost, chronicity or delayed recovery, and severity of the problem due to the individual's problematic musculoskeletal condition.
Fear-Avoidance Beliefs Questionnaire (FABQ) | Change from Baseline FABQ at 12 weeks
  The FABQ consists of 16 items and is divided into 2 subscales. The items are scored on a 7-point Likert scale (from strongly disagree to strongly agree). The score of each subscale is used independently. Higher scores represent more fear avoidance beliefs.
Oswestry Disability Index (ODI) | Change from Baseline ODI at 12 weeks
  The Oswestry Disability Index consists of 10 questions measuring functional status. Each question is evaluated between 0 and 5 points and the total maximum score is 50. Higher score indicates more disability.
Lumbar region proprioception measurement | Change from Baseline proprioception measurement at 12 weeks
  Subjects are asked to stand in a neutral position, with knees straight and weight equal to both feet. To measure lumbar repositioning errors in flexion, the first inclinometer is placed on the lateral chest (T12 level) and the second inclinometer on the hemipelvis (S1 level). The primary inclinometer (T12) and the secondary inclinometer (sacral midpoint) are used in the frontal plane to record the lateral bending angle error. Velcro straps are used to secure the digital inclinometer. The inclinometer is calibrated by the examiner to a starting position (0 degrees). Subjects memorize this neutral position for a few seconds, perform active full flexion and then return to the neutral position. Displacement accuracy is measured in degrees.
Five Times Sit to Stand Test (5TSST) | Change from Baseline 5TSST at 12 weeks
  A chair without armrests, with a 28.5 cm deep seat and backrest and adjustable height is used for the tests. Subjects start in a seated position, with their arms in the desired position and their backs against the chair backrest. The following verbal instructions are given: "Please stand up and sit down 5 times as quickly as possible. Straighten your knees when standing up and lean your back against the backrest when sitting down." Timing with the digital stopwatch is started manually with the instruction "Start" and stopped when the subject's back touches the backrest after the fifth standing up.
Timed Up and Go Test (TUG) | Change from Baseline TUG at 12 weeks
  Participants sit in a chair with arms, hips and knees bent approximately 90◦ and feet resting on the floor. Lower limb orthoses are worn if used. Participants are asked to stand up, walk 10 steps, walk around a mark on the floor, walk back to the chair and sit down. The timing of the TUG test starts with the standing movement after the "ready, go" signal and ends when the participants are seated in the chair and the movement is finished.

CONTACTS AND LOCATIONS:
Overall Officials: Fatih Özden, PhD, Principal Investigator — Muğla Sıtkı Koçman University
Locations (1):
- Muğla, Muğla, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No